CLINICAL TRIAL: NCT04156737
Title: A Comparative Clinical Evaluation of a New TECNIS® Presbyopia-correcting Intraocular Lens Against a Trifocal Intraocular Lens
Brief Title: A Comparative Study of TECNIS Symfony Plus IOL and a Trifocal IOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Surgical Vision, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SUR-IOL-652-3002
Record Dates: First submitted 2019-11-06; First posted 2019-11-07 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-08

CONDITIONS: Cataract; Refractive Error
MeSH Terms: conditions — Cataract; Refractive Errors

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Unmasked study personnel at the site will be trained to the randomization process through the EDC system and will randomize subjects. The surgeon and the operative staff will know which lens type is implanted. There may also be site coordinators and other site study staff, such as those performing slit-lamp exams, who will be unmasked. Unmasked study site staff will be instructed not to disclose the lens type the subject received or to talk about the lens to any masked evaluators or to the study subjects. The subjects and the study technicians performing the postoperative vision tests are to be masked through study completion. To maintain subject masking, a temporary IOL implant identification card will be issued to the subject at the time of surgery. Following completion of the final study exam, each subject will be given the permanent IOL implant identification card.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Investigational Lens (Experimental): TECNIS Symfony plus IOL Model ZHR00V
  Interventions: Device: TECNIS Symfony plus IOL Model ZHR00V
- Control Lens (Active Comparator): Trifocal Intraocular Lens
  Interventions: Device: Trifocal Intraocular lens

INTERVENTIONS:
Device: TECNIS Symfony plus IOL Model ZHR00V — IOL replaces the natural lens removed during cataract surgery
  Arms: Investigational Lens
Device: Trifocal Intraocular lens — IOL replaces the natural lens removed during cataract surgery
  Arms: Control Lens

SUMMARY:
This is a multicenter, prospective, randomized, subject- and evaluator-masked, bilateral-implant study conducted at up to 15 sites worldwide. A total of up to 280 subjects will be randomized in a 1:1 ratio for implantation with either the TECNIS Symfony plus IOL Model ZHR00V or the Trifocal IOL. This will ensure that data from at least 100 subjects in the TECNIS Symfony plus lens group and at least 100 subjects in the Trifocal lens group will be available for analysis at the 6-month follow-up timepoint. All subjects will be followed for up to 6 months postoperative.

ELIGIBILITY:
Inclusion Criteria:

(all criteria apply to both eyes):

* Age 22 and older
* Bilateral cataracts or clear crystalline lenses for which posterior chamber IOL implantation has been planned
* Potential postoperative best corrected distance visual acuity (BCDVA) of 0.66 decimal (20/30 or 6/9 Snellen) or better
* Predicted postoperative corneal astigmatism less than 1.0 D, including posterior corneal astigmatism (PCA)
* Clear intraocular media other than cataract in each eye
* Availability, willingness and sufficient cognitive awareness to comply with examination procedures
* Ability to understand, read, and write English or the local language in which the informed consent and questionnaires are provided
* Written informed consent for participation in the study and data protection.

Exclusion Criteria:

* (including device labeling, all criteria apply to both eyes):

  * Require an intraocular lens power outside the available range of +14.0 to +26.0 D
  * Irregular corneal astigmatism (as evaluated by topography)
  * Prior corneal refractive (LASIK, LASEK, RK, PRK, etc.) or intraocular surgery, including prophylactic peripheral iridotomies and peripheral laser retinal repairs
  * Corneal abnormalities such as stromal, epithelial or endothelial dystrophies (e.g., any observed guttata) that are predicted to cause visual acuity loss to a level worse than 0.66 decimal (20/30 or 6/9 Snellen) during the study
  * Inability to achieve keratometric stability for contact lens wearers
  * Recent ocular trauma or ocular surgery that is not resolved/stable or may affect visual outcomes or increase risk to the subject
  * Pupil abnormalities that may affect visual outcomes or increase risk to the subject
  * Subjects with diagnosed degenerative visual disorders (e.g., macular degeneration or other retinal disorders) that are predicted to cause visual acuity loss to a level worse than 0.66 decimal (20/30 or 6/9 Snellen) during the study
  * Subjects with conditions associated with increased risk of zonular rupture, including capsular or zonular abnormalities that may lead to IOL decentration or tilt, such as pseudoexfoliation, trauma, or posterior capsule defects
  * Use of systemic or ocular medications that, in the opinion of the investigator, may affect vision
  * Prior, current, or anticipated use during the 6-month study of tamsulosin or silodosin that may, in the opinion of the investigator, confound the outcome or increase the risk to the subject (e.g., poor dilation or a lack of adequate iris structure to perform standard cataract surgery)
  * Poorly-controlled diabetes or hypertension that, in the opinion of the investigator, may mpact visual outcome or increase the risk to the subject
  * Acute, chronic, or uncontrolled systemic or ocular disease or illness that, in the opinion of the investigator, would increase the operative risk or confound the outcome(s) of the study (e.g., immunocompromised, connective tissue disease, suspected glaucoma, glaucomatous changes in the fundus or visual field, ocular inflammation, etc.). Note: controlled ocular hypertension without glaucomatous changes (optic nerve cupping and visual field loss) is acceptable.
  * Known ocular disease or pathology that, in the opinion of the investigator,

    * may affect visual acuity (e.g., ocular surface conditions)
    * may require surgical intervention during the study (macular degeneration, cystoid macular edema, diabetic retinopathy, uncontrolled glaucoma, etc.)
    * may be expected to require retinal laser treatment or other surgical intervention during the study (macular degeneration, cystoid macular edema, diabetic retinopathy, etc.)
  * Pregnancy, planned pregnancy, presently lactating, or another condition associated with hormonal fluctuation that could lead to refractive changes
  * Concurrent participation or participation within 60 days prior to the preoperative visit in any other clinical trial
  * Desire for monovision correction

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2020-01-24 (Actual); Primary Completion 2021-07-14 (Actual); Study Completion 2021-07-14 (Actual)

PRIMARY OUTCOMES:
Binocular distance-corrected VA of 20/25 | 3 months
  Percent of subjects who achieve binocular distance-corrected VA of 20/25 (6.7.5) Snellen or better at far, intermediate, and near (40 cm)
Binocular uncorrected VA of 20/32 | 3 months
  Percent of subjects who achieve binocular uncorrected VA of 20/32 or better at far and near (40 cm)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Surgical Vision Clinical Trials, Study Director — Johnson & Johnson Surgical Vision
Locations (5):
- Auckland Eye Institute, Remuera, Auckland, New Zealand
- Asian Eye Institute, Makati, Philippines
- Spain (3):
  - Clinica de Oftalmologia de Cordoba, Córdoba
  - Centro Ocular de Alta Technologia Oftalmos, Madrid
  - Miranza IOL Madrid, Madrid

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Devices Companies have an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA project site at http://yoda.yale.edu
URL: http://yoda.yale.edu/